CLINICAL TRIAL: NCT00679315
Title: Efficacy and Safety of Alfuzosin for the Treatment of Non-neurogenic Voiding Dysfunction in Female: An 8 Week Prospective, Randomized Double Blind, Placebo-Controlled, Parallel Group Study (Phase Ⅱ)
Brief Title: Efficacy and Safety of Alfuzosin for the Treatment of Voiding Dysfunction in Female
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Handok Inc. (Industry); The Korean Urological Association (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-07-073
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Voiding Dysfunction
Keywords: female voiding dysfunction; alpha adrenoreceptor antagonists; IPSS or American Urological Association symptom index
MeSH Terms: interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpha blocker (Experimental): alfuzosin hydrochloride XL 10mg
  Interventions: Drug: alfuzosin hydrochloride XL 10mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alfuzosin hydrochloride XL 10mg — One tablet to be taken daily after a meal before bedtime for 8 weeks.
  Other Names: Xatral® XL
  Arms: Alpha blocker
Drug: Placebo — One tablet to be taken daily after a meal before bedtime for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore the efficacy of Alfuzosin (10 mg, qd) in reducing the score of International Prostate Symptom Score (IPSS) from baseline to 8 weeks of treatment in female patients with voiding dysfunction.

DETAILED DESCRIPTION:
Trial design

Phase II, multi-center, randomized, double-blind, placebo-controlled, parallel group study to evaluate the clinical efficacy and safety of alfuzosin (10mg, qd) from baseline to 8 weeks of treatment in female patients with non-neurogenic voiding dysfunction.

Efficacy Assessment

1. Primary efficacy endpoint

   Actual change in the score of IPSS from baseline to 8 weeks of treatment.
2. Secondary efficacy endpoint

   * IPSS parameters
   * Percent change in the score of IPSS from baseline to 4 and 8 weeks of treatment.
   * Actual and percent changes in the sub-scale of IPSS from baseline to 4 and 8 weeks of treatment
   * Storage score: sum of questions 2, 4 and 7
   * Voiding score: sum of questions 1, 3, 5 and 6
   * Scored form of the Bristol Female Lower Urinary Tract Symptoms (BFLUTS-SF)parameters
   * Actual and Percent change in BFLUTS-SF from baseline to 4 and 8 weeks of treatment.
   * Actual and percent changes in the sub-scale of BFLUTS-SF from baseline to 4 and 8 weeks of treatment

     * BFLUTS-FS: sum scores F1-F4
     * BFLUTS-VS: sum scores V1-V3
     * BFLUTS-IS: sum scores I1-I5
     * BFLUTS-sex: sum scores S1 & S2
   * Uroflowmetry & PVR parameters

     * Numeric and percent changes from baseline to 4 and 8 weeks of treatment.
     * Maximum flow rate (mL/s)
     * Average flow rate (mL/s)
     * Post-void residual urine (mL)
     * Micturition diary parameters
     * Change in mean number of micturitions per 24 hours at weeks 4 and 8 relative to baseline
     * Percent change of micturitions per 24 hours at weeks 4 and 8 relative to baseline
     * Change in mean number of nighttime micturitions per 24 hours at weeks 4 and 8 relative to baseline
     * Percent change of nighttime micturitions per 24 hours at weeks 4 and 8 relative to baseline
     * Change in mean number of urgency episodes per 24 hours at weeks 4 and 8 relative to baseline (Urgency episodes are defined as those with Bladder Sensation Scale rating of ≥ 3 in the diary).
     * Percent change of urgency episodes per 24 hours at weeks 4 and 8 relative to baseline
     * Change in the mean and sum rating on the Bladder Sensation Scale at weeks 4 and 8 relative to baseline
     * Quality of life (QoL) parameters
     * Change in Bother score of IPSS from baseline to 4 and 8 weeks of treatment.
     * Change in QOL subscale scores of BFLUTS SF from baseline to 4 and 8 weeks of treatment
     * BFLUTS-QoL: Sum scores QoL1-QoL5
     * Patient Perception of Bladder Condition (PPBC)
     * Change from baseline in PPBC after 8 weeks of double-blind treatment
     * Benefit, Satisfaction, and Willingness to Continue (BSW) Questions
     * Patient Perception of Treatment Benefit at week 8
     * Patient Perception of Treatment Satisfaction at week 8
     * Willingness to continue with treatment at week 8

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 18
* Have voiding symptoms as chief complaints over 3 months
* IPSS symptom score ≥ 15
* A peak flow rate <12 mL/sec with a minimum voided volume of 100 mL and/or a postvoid residual urine volume >150 mL
* Underwent pressure-flow study

Exclusion Criteria:

* Patients who meet any of the following criteria are to be excluded from the study:
* Neurogenic voiding dysfunction
* Anatomic causes of bladder outlet obstruction
* Perform physical examination in patients diagnosed as BOO in pressure-flow study by urethral evaluation with 16 Fr urethral sound: if there is resistance to 16Fr sound, it will be diagnosed as anatomical BOO and the patients can not participate in the study.
* Previous surgical procedures related to incontinence or cystocele
* Pregnant or nursing women
* Intake of medications and drugs affecting bladder function: alpha blocker, anticholinergic
* Anticholinergic drugs: Tolterodine, Oxybutynin, Propiverin, Trospium, Solifenacin, SSRI including TCA
* Cholinergic drug: Bethanechol
* Any other blocker other than alfuzosin
* patients can be enrolled after wash-out
* Any positive urine culture had to be successfully treated before the recruitment.
* Clinically significant ( ≥ Stamey grade II/III) stress incontinence as determined by the investigator and confirmed for female patients by a cough provocation test.
* Recurrent UTIs defined as having been treated for symptomatic UTIs ≥ 4 times in the last year
* Diagnosed or suspected interstitial cystitis
* Patients with marked cystocele or other clinically significant pelvic prolapse.
* Treatment within the 14 days preceding randomization, or expected to initiate treatment during the study with:
* Estrogen treatment started more than 2 months prior to inclusion will be allowed
* Receipt of any electrostimulation or bladder training within the 14 days before randomization, or expected to start such treatment during the study.
* Hypersensitive to the study drug
* Orthotopic hypotension or history of orthotopic hypotension
* Intake of calcium channel blockers
* Severe hepatic or renal dysfunctions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Actual change in the score of IPSS from baseline to 8 weeks of treatment. | 8 weeks of treatment

SECONDARY OUTCOMES:
IPSS parameters | 4 and 8 weeks of treatment.
BFLUTS-SF parameters | 4 and 8 weeks of treatment
Uroflowmetry & PVR parameters | 4 and 8 weeks of treatment
Micturition diary parameters | 4 and 8 weeks of treatment
Quality of life parameters | 4 and 8 weeks of treatment
Patient Perception of Bladder Condition | 8 weeks of treatment
Benefit, Satisfaction, and Willingness to Continue (BSW) Questions | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (9):
- South Korea (9):
  - Samsung Medical Center, Seoul, Seoul
  - Chungnam National University Hospital, Daejeon
  - Holy Family Hospital, The Catholic University of Korea, Kyonggi-do
  - Pusan National University Hospital, Pusan
  - Cheil General Hospital & Women's Healthcare Center, College of Medicine, Kwandong University, Seoul
  - Seoul National University Hospital, Seoul
  - Anam Hospital, College of Medicine, Korea University, Seoul
  - Kangnam St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Asan Medical Center, Ulsan College of Medicine, Seoul